CLINICAL TRIAL: NCT04995952
Title: Comparison Of Gross Motor Task Training And Trunk Targeted Training On Balance, Range Of Motion And Community Participation In Children With Cerebral Palsy
Brief Title: Comparsion of Gross Motor Task Training and Trunk Trageted Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: khadija liaquat (Other)
Responsible Party: Sponsor-Investigator, khadija liaquat, senior lecturer, Riphah International University
Organization: Riphah International University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RiphahIU maryam
Record Dates: First submitted 2021-08-06; First posted 2021-08-09 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Cerebral Palsy
Keywords: Cerebral plasy; Trunk targeted training; Gross motor trageted training; Balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gross motor training activity (Experimental): Gross motor training activity It includes training of motor components of child grossly
  Interventions: Behavioral: Gross motor training
- Trunk targeted training (Experimental): In this training group the particpiants were given the exercises that were focused the truck muscles
  Interventions: Behavioral: Trunk targeted training

INTERVENTIONS:
Behavioral: Gross motor training — Gross motor training activity (1 hour session, 3 times a week for 3 months). Pre ad post assessments will be taken. The Gross motor training activity will include: sit to stand, step-ups and walking. The sit to stand will be performed for 20 minutes involving 20 repetitions. We will progress from high seat sit to stand to low seat sit to stand. The step up will progress initially from a bench having low height to high height and then to stepping of stairs for 20 minutes involving 30 repetitions. The walking will occur from 3m walk and then increasing the distance
  Arms: Gross motor training activity
Behavioral: Trunk targeted training — Trunk targeted training (1hour session, 3 times a week for 3 months). Pre and Post assessment will be evaluated. The trunk targeted training will include: weight supported treadmill walk, specific trunk exercises with vibration therapy and reaching forward to the limits of stability.
  Specific trunk exercises will involve stride sitting to standing, sitting on a roll and moving the roll in diagonal and forward backward directions along with giving vibrational therapy on wobble board, side sitting. This activity will be performed for 30 minutes with 30 repetitions. Reaching forward to the limits of stability exercises will be performed. Asking the children to hold objects from right hand while reaching for an object on left side and vice versa. This will be performed for 20 minutes having 20 repetitions.
  Arms: Trunk targeted training

SUMMARY:
In this study trunk, targeted training and gross motor function training were compared their effect on functional status, range of motion, and community participation of cerebral palsy children

DETAILED DESCRIPTION:
In this project a randomized clinical trial was be conducted to determine the comparison of gross motor training technique and trunk training therapy on balance, Range of motion and community participation in children with diplegic cerebral palsy. This study aim to compare the effects of both the treatments to improve balance, quality of life and community participation. The sample was being collected according to inclusion and exclusion criteria using a convenient sampling technique within period of 6 months. The participants were be randomly allocated in two groups' .Group A received gross motor training which included sit to stand, step up and walking for 1 hour/day/3 days a week for 3 months. Group B received trunk targeted training for 1 hour/day/3 days a week for 3 months which included treadmill walking, reaching forward to the limits of stability and specific truncal activities with vibration and proprioception. The post treatment assessments was done via early assessment of balance, goniometer, and functional mobility assessment

ELIGIBILITY:
Inclusion Criteria male & female.

* GMFCS III V
* Age 8to12 years
* Diplegic cerebral palsy
* Hypoxic brain injury
* Diagnosed with a gross motor delay by the pediatrician.

Exclusion Criteria:

* Children having a cognitive or psychiatric disorder.
* Children with known congenital limb anomaly
* Children with some chromosomal defect

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Functional mobility assessment | 10 minutes
  It classifies the functional mobility of children between ages 4-18 years of age with cerebral palsy. The scale can be used to classify children's functional mobility, document change over time in the same child and to document change. The FMS rates walking ability at three specific distances, 5, 50 and 500 meters, (or 5, 50, 500 yards). This represents the child's mobility in the home, at school and in the community setting
Pediatric Berg Balance Scale | 20 minutes
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children and children with cerebral palsy. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
Goniometer | 10 minutes
  This is an instrument which is used to measure the range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Prof S Shakil Ur Rehman, Phd, Study Director — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No